CLINICAL TRIAL: NCT02209688
Title: Administration of ESR 1150 CL in Ascending Doses of 0.5, 1, 2, 4 and 8 mg in an Open, Group Comparison and Placebo-controlled Design (Placebo Randomised Double Blind in the Dose Groups) for the Assessment of Safety, Tolerability (Maximum Tolerated Dose, MTD), Pharmacokinetics and Pharmacodynamics in 5 Groups of 8 Female and 5 Male Healthy Subjects, and 4 mg Additionally in Fed State, in a Cross Over Design. Safety, Tolerability and Pharmacokinetics of MTD/4, MTD/2 and MTD in 6 Healthy Male Subjects, Identified as CYP2D6 and/or "Spartein" Poor Metabolizers, in a 3-fold Cross Over, Open Study.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ESR 1150 CL in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1172.2
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (3):
- ESR 1150 CL dose escalation fasted (Experimental)
  Interventions: Drug: ESR 1150 CL
- ESR 1150 CL fed (Experimental)
  Interventions: Drug: ESR 1150 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESR 1150 CL
  Arms: ESR 1150 CL dose escalation fasted; ESR 1150 CL fed
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study was to obtain safety and tolerability data and first pharmacokinetic and pharmacodynamic data of escalating doses of ESR 1150 CL.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Caucasian subjects as determined by results of screening
* Written informed consent in accordance with Good Clinical Practice and local legislation given
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20 % and ≤ + 20 %
* for first part of study: extensive metabolizers of CYP2D6 and/or "spartein" type; for second part of study: poor metabolizers of CYP2D6 and/or "spartein"

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders of neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (≤ 1 month prior to administration or during the trial, except for oral contraceptives)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial except for oral contraceptives)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/days)
* Drug abuse
* Blood donation > 100 ml (≤ 4 weeks prior to administration or during the trial)
* Excessive physical activities (≤ 10 days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* Females only:

  * No reliable contraception (examples of reliable contraception: oral contraceptives, 3-month injection, intrauterine device, sterilisation, condoms + spermicide)
  * pregnancy or breast feeding period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2000-02; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 30 days
Area under the curve (AUC) | up to 24 hours after administration
Maximum concentration (Cmax) | up to 24 hours after administration
Time to maximum concentration (tmax) | up to 24 hours after administration
Apparent total plasma clearance (CLtot/f) | up to 24 hours after administration
Apparent volume of distribution (Vz/f) | up to 24 hours after administration
Elimination half-life (t1/2) | up to 24 hours after administration
Amount excreted in urine (Ae) | up to 24 hours after administration
Maximum flow rate (Qmax) | up to 8 hours after administration
  assessed by free uroflowmetry
Average flow rate (Qave) | up to 8 hours after administration
  assessed by free uroflowmetry
Voided volume (Vcomp) | up to 8 hours after administration
  assessed by free uroflowmetry
Voiding time (T100) | up to 8 hours after administration
  assessed by free uroflowmetry
Time to maximum flow (TQmax) | up to 8 hours after administration
  assessed by free uroflowmetry
Residual urinary volume | up to 8 hours after administration
  assessed by means of transabdominal ultrasound evaluation
Assessment of micturition pattern | up to 8 hours after administration
  evaluated by Independent reviewer
Amount of inhibition constants (Ki) at α1A, adrenoreceptor subtype level | up to 8 hours after administration
  assessed by ex vivo radioreceptor assay